CLINICAL TRIAL: NCT00362206
Title: A Multicenter, Double-Blind, Randomized, Forced-Titration Study to Compare the Efficacy and Safety of the Combination of 145 mg Fenofibrate and 20 or 40 mg Simvastatin With 40 mg Pravastatin Monotherapy in Patients With Mixed Dyslipidemia at Risk of Cardiovascular Disease Not Adequately Controlled by 40 mg Pravastatin Alone
Brief Title: Comparison of the Combination of Fenofibrate and Simvastatin Versus Pravastatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Martine Guy, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C LF0242780-01 05 04; 2006-000515-15
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Hyperlipidemia
Keywords: Hyperlipidemia Combined, efficacy combination fenofibrate simvastatin versus pravastatin; Hyperlipidemia Combined
MeSH Terms: conditions — Hyperlipidemias | interventions — Fenofibrate; Simvastatin; Pravastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Fenofibrate/Simvastatin
- 2 (Experimental)
  Interventions: Drug: Fenofibrate/Simvastatin
- 3 (Active Comparator)
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Fenofibrate/Simvastatin — Combination of Fenofibrate and Simvastatin 20mg
  Arms: 1
Drug: Fenofibrate/Simvastatin — Combination of Fenofibrate and Simvastatin 40 mg
  Arms: 2
Drug: Pravastatin — Pravastatin 40 mg
  Arms: 3

SUMMARY:
Mixed or combined hyperlipidemia is a common metabolic disorder characterized by both hypercholesterolemia and hypertriglyceridemia. Statins and fibrates have complementary mechanisms and can be coadministered to patients with mixed hyperlipidemia.The overall objective of the study is to compare the efficacy and safety of combining fenofibrate and simvastatin versus pravastatin monotherapy in patients with mixed hyperlipidemia at risk of cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Mixed dyslipidemia

Exclusion Criteria:

* Known hypersensitivity to fenofibrates or simvastatin or pravastatin
* Pregnant or lactating women
* Contra-indication to fenofibrate or simvastatin or pravastatin
* Unstable or severe cardiac disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to 12 weeks of treatment in Triglycerides | 12 weeks
Percent change from baseline to 12 weeks of treatment in HDL-C | 12 weeks
Percent change from baseline to 12 weeks of treatment in LDL-C | 12 weeks

SECONDARY OUTCOMES:
Percent change from baseline to 12 weeks of treatment in Triglycerides | 24 weeks
Percent change from baseline to 12 weeks of treatment in HDL-C | 24 weeks
Percent change from baseline to 12 weeks of treatment in LDL-C | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (41):
- Greece (3):
  - Site 40, Athens
  - Site 39, Ioannina
  - Site 41, Thessaloniki
- Israel (10):
  - Site 37, Beer Yaakov
  - Site 19, Haifa
  - Site 22, Holon
  - Site 18, Jerusalem
  - Site 38, Kfar Saba
  - Site 17, Ramat Gan
  - Site 21, Ramat Gan
  - Site 20, Rehovot
  - Site 24, Safed
  - Site 23, Tel Aviv
- Romania (7):
  - Site 5, Arad
  - Site 7, Bacau
  - Site 1, Bucharest
  - Site 6, Cluj-Napoca
  - Site 4, Oradea
  - Site 3, Ploieşti
  - Site 2, Târgu Mureş
- Russia (8):
  - Site 27, Barnaul
  - Site 31, Kemerovo
  - Site 32, Krasnoyarsk
  - Site 25, Moscow
  - Site 28, Novosibirsk
  - Site 29, Saint Petersburg
  - Site 26, Smolensk
  - Site 30, Voronezh
- South Africa (13):
  - Site 10, Alberton
  - Site 9, Bloemfontein
  - Site 14, Cape Town
  - Site 35, Durban
  - Site 36, eMkhomazi
  - Site 33, Hillcrest
  - Site 34, Kempton Park
  - Site 16, Komatipoort
  - Site 13, Krugersdorp
  - Site 11, Parow
  - Site 12, Port Elizabeth
  - Site 8, Pretoria
  - Site 15, Worcester